CLINICAL TRIAL: NCT07090057
Title: The Effect of Targeting the Plantaris Muscle-tendon Unit in Surgical Correction of Ankle Equinus in Children
Brief Title: The Effect of Targeting the Plantaris Muscle-tendon in Surgical Correction of Ankle Equinus in Children
Acronym: Plantaris Sx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00123505
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Toe Walking; Cerebral Palsy; Hereditary Spastic Paraparesis; Traumatic Brain Injury; Spinal Cord Injury; Spinal Cord Tethering; Stroke; Hereditary Sensory-motor Neuropathy
Keywords: tendoachilles lengthening; gastrocnemius recession; Plantaris lengthening
MeSH Terms: conditions — Cerebral Palsy; Spastic Paraplegia, Hereditary; Brain Injuries, Traumatic; Spinal Cord Injuries; Stroke; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Intervention Model Description: Data will be collected from 42 children undergoing surgical intervention for ankle equinus. Subjects will be randomly allocated into two groups of equal size: 1) plantaris lengthened before the lengthening of gastrocsoleus and 2) plantaris lengthened after gastrocsoleus lengthening. All surgical procedures for each patient will be completed in a single setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tendoachilles (TA) lengthening or gastrocnemius (GN) recession, then Plantaris tenotomy (Experimental): Participants undergo Tendoachilles (TA) lengthening or gastrocnemius (GN) recession surgery before Plantaris tenotomy.
  Interventions: Procedure: Tendoachilles (TA) lengthening or gastrocnemius (GN) recession, then Plantaris tenotomy
- Plantaris tenotomy, then Tendoachilles (TA) lengthening or gastrocnemius (GN) recession (Experimental): Participants undergo Plantaris tenotomy surgery before Tendoachilles (TA) lengthening or gastrocnemius (GN) recession.
  Interventions: Procedure: Plantaris tenotomy, then Tendoachilles (TA) lengthening or gastrocnemius (GN) recession

INTERVENTIONS:
Procedure: Tendoachilles (TA) lengthening or gastrocnemius (GN) recession, then Plantaris tenotomy — Participants undergo Tendoachilles (TA) lengthening or gastrocnemius (GN) recession surgery before Plantaris tenotomy.
  Arms: Tendoachilles (TA) lengthening or gastrocnemius (GN) recession, then Plantaris tenotomy
Procedure: Plantaris tenotomy, then Tendoachilles (TA) lengthening or gastrocnemius (GN) recession — Participants undergo plantaris tenotomy surgery before Tendoachilles (TA) lengthening or gastrocnemius (GN) recession.
  Arms: Plantaris tenotomy, then Tendoachilles (TA) lengthening or gastrocnemius (GN) recession

SUMMARY:
Tight ankle muscles can produce ankle equinus (limited ability to pull the foot upward) and occur often in children, significantly impacting their ability to walk. If not treated, children with ankle equinus frequently experience reduced function and long-term foot problems, such as pain. Currently, treatment options include surgery or Botulinum toxin (BoNTA) injection into the large calf muscles that point the foot downwards, aiming to reduce their tightness. However, these treatments can be less effective over time, can create prolonged calf weakness, and may require long-term bracing. Another small muscle in the leg, the plantaris, is believed to have some contribution to equinus in many children. It is sometimes included in treatment plans for equinus but its contribution is poorly understood. It is unclear whether targeting the plantaris alone could lead to better treatment of ankle equinus. Understanding the effect of treatments targeting the plantaris could help clinicians improve the management of ankle equinus.

In this study, the investigators will look at the impact of surgical treatment to the plantaris in ankle equinus. The investigators hypothesize that the plantaris is a significant contributor to equinus.

In this study, data will be collected from children undergoing surgical correction of ankle equinus, including lengthening of the plantaris and lengthening of the larger muscles producing equinus (the gastrocsoleus mechanism). Children will be randomly assigned to have either their plantaris or the gastrocsoleus lengthening be done first during surgery. All children will have both structures lengthened during surgery, only the order will be varied and all surgical procedures for each patient will be completed in a single setting. In both groups, maximum passive ankle dorsiflexion (upwards bend of the ankle with the knee straight) will be measured before and after each structure is lengthened. The outcome is maximum passive ankle dorsiflexion (upwards bend of the ankle) with the knee straight.

The investigators expect that maximum passive ankle dorsiflexion will increase after lengthening of the plantaris. Understanding the contribution of the plantaris muscle in ankle equinus could lead to significant improvements in the treatment of children with tight ankles.

DETAILED DESCRIPTION:
Children demonstrating equinus gait, characterized as <10° of ankle dorsiflexion relative to the leg, are commonly referred for specialist assessment. Equinus gait or deformity can occur in isolation (e.g. idiopathic toe-walking), with other foot deformities (e.g. clubfoot), or with underlying neuromotor conditions (e.g. cerebral palsy). A 2019 study found 83.3% of patients surveyed with cerebral palsy had equinus.

In children with underlying spasticity and no significant contracture, chemodenervation via Botulinum toxin (BoNTA) injections of the gastroc-soleus (GS) complex is often used to maintain functional range and optimize gait. Typically, injections become less effective over time, often leading to equinus contracture, functional impairment, and the need for orthoses or surgery. Once surgical intervention (i.e. tendoachilles (TA) lengthening or gastrocnemius (GN) recession) is required, contracture of the plantaris muscle has also been noted, usually requiring concomitant or later lengthening via tenotomy. Surgical GS lengthenings to treat ankle equinus can result in prolonged and sometimes incomplete recovery of ankle plantarflexion strength despite intensive physiotherapy, adversely affecting gait and lower limb function.

The presence and course of plantaris are believed to be variable. Recent evidence indicates that it is present in 98-100% of the population while historical estimates ranged from 80-93%. Historically considered a vestigial structure with no significant functional impact, more recently, plantaris contraction is considered to impact knee flexion and ankle plantarflexion as well as possibly contribute to external rotation of the lower leg and hindfoot inversion, similar to the GN. Given these potential functional similarities and empiric intra-operative observations of improved ankle dorsiflexion with plantaris lengthening in addition to GS complex lengthening, a plantaris tenotomy is often performed during surgery for equinus contracture. However, clinical recognition of the plantaris contribution to equinus gait and/or contracture remains inconsistent, and the effect of treatments targeting the plantaris are not well described in the literature.

The overall goal of this proposed study is to examine the contribution of the plantaris to ankle equinus by assessing the short-term impact of surgical treatment targeting the plantaris muscle-tendon unit to manage children with equinus gait and/or contracture.

The trial will compare changes to passive ankle dorsiflexion after plantaris tenotomy performed either a) before TA lengthening or GN recession or b) after TA lengthening or GN recession (in a single surgical encounter).

If this surgical trial finds that plantaris significantly contributes to equinus contracture, it may support using exclusively open surgical techniques (rather than percutaneous), so the plantaris can be identified and addressed adequately. In addition, if the effect of plantaris is significant, it is possible that early isolated release of the plantaris tendon may be a treatment option while preserving the gastrocsoleus complex and thereby reducing post-operative weakness. This approach would benefit from the development of minimally invasive techniques to identify the tendon but has the potential reduce the long-term requirement for Achilles tendon lengthening with improved preservation of plantarflexion strength by reducing the feedback mechanism from the plantaris to the gastrocsoleus complex.

The investigators hypothesize that the plantaris significantly contributes to equinus contracture in children and that plantaris tenotomy in this population significantly improves passive ankle dorsiflexion, independent of the GS mechanism.

The primary objectives of this study are to:

1) Compare the effect of plantaris tenotomy in the setting of equinus contracture on passive ankle dorsiflexion relative to that of TA lengthening or GN recession.

The secondary objectives are to:

1. Quantify the proportion of participants with an identifiable plantaris
2. Describe the location of the insertion of the plantaris tendon in those with an identified plantaris

This is a single-centre, randomized intra-operative clinical study involving pediatric patients undergoing surgery for equinus contracture at the Stollery Children's Hospital. All procedures will occur within a single operative session and will be performed by pediatric orthopedic surgeons. Pre- and post-intervention assessments will be performed intra-operatively, so minimal loss to follow-up is expected. Maximum passive ankle dorsiflexion will be measured by the surgeon with a sterile goniometer at four different time points (before and after lengthening of each tendon/aponeurosis), with the knee maximally extended. To minimize confounding by any co-existing intrinsic foot deformities, ankle dorsiflexion will be measured with the long axis of the leg and long axis of the heel pad as the points of reference.

After both structures (i.e., plantaris tendon and GN aponeurosis or Achilles tendon) have been identified, the plantaris location will be documented. In GN recession cases where there is inadequate dorsiflexion after both procedures, the surgeon may complete a partial lengthening of the soleus at their discretion, with a fifth set of measurements documented after completion.

The study population will include children undergoing surgical lengthening of the GN or TA. 42 participants (21 per group, 20 for power and one in case a patient doesn't have a plantaris or whose physical examination changes between consent and surgery) will be included.

Due to the paucity of literature, estimate of required sample size is based on a minimal clinically important difference (MCID) derived from the experience of the study surgeons. There were 27 and 28 eligible patients in 2020 and 2021 respectively.

A member of the patient's care team (i.e. surgeon, nurse, or resident) will identify potential participants, completing a Consent to Contact from when patients are consented or scheduled for the index procedure. A Research Associate will contact the potential participant or their legal guardian and explain the study. If the potential participants wish to take part, they will provide consent via e-consent on REDCap. Once consent is obtained, notification will be sent to the treating surgeons' office, along with the participant's randomization allocation.

A computer-generated, uneven block randomization sequence will be used to randomize participants to one of the two groups.

Descriptive statistics will characterize baseline demographics and any systematic differences among groups will be risk-adjusted. Maximum passive ankle dorsiflexion during surgery will be examined using ANOVA or corresponding Kruskal-Wallis model.

Summary:

Surgery is routinely done for patients with equinus contracture involving lengthening of the tendoachilles or gastrocnemius and then plantaris to achieve the desired ankle range of motion. In this study, the investigators want to understand the contribution of plantaris to ankle equinus in children. In the future, if plantaris can be cut first and the desired range of motion is obtained, then the tendoachilles and gastrocnemius need not be cut. This will dramatically reduce post-operative recovery time and will likely preserve ankle plantarflexor strength.

ELIGIBILITY:
Inclusion Criteria (All of the following criteria must be met):

* Ability to provided informed consent/assent in English.
* Pediatric patients (4-17 years) who have consented for surgery for the management of equinus contracture * (either TA lengthening or GN recession) at the Stollery Children's Hospital
* Known underlying diagnosis of any of the following: idiopathic toe walking, cerebral palsy, hereditary spastic paraparesis, traumatic brain injury, spinal cord injury/tethering, hereditary sensory-motor neuropathy, stroke
* Ability to maintain hindfoot and midfoot neutral during assessment
* Passive plantarflexion on affected side greater than 20° and greater than degree of equinus contracture.

  * Note: may be isolated or in conjunction with other orthopaedic procedures; in bilateral ankle equinus procedures, data will be collected bilaterally, but included as a single participant (i.e., single randomization).

Exclusion Criteria (Any one or more of the following):

* Unable to provide informed consent/assent in English.
* Previous surgery for equinus
* Limb deficiency on affected side
* Knee flexion contracture of greater than 5°
* Surgical intervention of the lower extremities below the affected knee in the last twelve months
* BoNTA injections below the affected knee within the last six months
* Known or suspected arthrofibrosis.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum passive ankle dorsiflexion | Prior to skin incision
  Ankle dorsiflexion (unit: degree) will be measured by the surgeon with a sterile goniometer during the surgery.
Maximum passive ankle dorsiflexion | Prior to division of first tendon/aponeurosis
  Ankle dorsiflexion (unit: degree) will be measured by the surgeon with a sterile goniometer during the surgery.
Maximum passive ankle dorsiflexion | After division of first tendon/aponeurosis
  Ankle dorsiflexion (unit: degree) will be measured by the surgeon with a sterile goniometer during the surgery.
Maximum passive ankle dorsiflexion | After division of second tendon/aponeurosis
  Ankle dorsiflexion (unit: degree) will be measured by the surgeon with a sterile goniometer during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sukhdeep Dulai, MD, MHSc, FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No